| Division | • | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | • | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A three part, non-randomised, open label study designed to assess the pharmacokinetics of GSK2982772 following administration of minitab modified release formulations in capsule relative to an immediate release reference tablet formulation (Part A), the pharmacokinetics of escalating, repeat doses of a selected minitab modified release prototype (Part B) in healthy subjects, and the pharmacokinetics of GSK2982772 following administration of modified release tablet formulations in the fed and fasted state (Part C) in healthy participants. |
|---|---|---|
| <b>Compound Number</b> | : | GSK2982772 |
| Effective Date | : | 24-JAN-2019 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205017.
- This RAP is intended to describe the PK, safety and tolerability analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Statistician (II Clinical Statistics) | 24-JAN-2019 | Email |
| Principal Statistician (II Clinical Statistics) | 23-JAN-2019 | Email |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development Manager (GCSD) | 23-JAN-2019 | Email |
| Clinical Development Director, Discovery<br>Medicine | 23-JAN-2019 | Email |
| Director (CPMS) | 23-JAN-2019 | Email |
| Project Physician Lead, iiTA | 23-JAN-2019 | Email |
| Senior Medical Director, GCSP SERM | 23-JAN-2019 | Email |
| Principal Data Manager (GCDO) | 23-JAN-2019 | Email |
| Principal Programmer (iiTA R&D PCPS) | 23-JAN-2019 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Senior Statistics Director (II Clinical Statistics) | 24-JAN-2019 | e-Signature |
| Programming Manager (II Clinical Programming) | 24-JAN-2019 | e-Signature |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DDUCTIO | ON | 6 |
| 2. | CLIMAN | | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | | |
| | | Change | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study C | Objective(s) and Endpoint(s) | 0 |
| | 2.3. | Study L | Design | ŏ |
| | 2.4. | Statistic | cal Hypotheses / Statistical Analyses | 9 |
| 3. | PI AN | NED AN | ALYSES | 10 |
| Ο. | 3.1. | | Analyses | |
| | 3.2. | | nalyses | |
| | 0.2. | i iiidi 7 ti | lary 500 | |
| 4. | ANAL <sup>*</sup> | YSIS PO | PULATIONS | 11 |
| | 4.1. | Protoco | ol Deviations | 11 |
| 5. | | | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | ENTION | IS | 12 |
| | 5.1. | Study T | reatment & Sub-group Display Descriptors | 12 |
| | 5.2. | | e Definitions | 13 |
| | 5.3. | | Considerations for Data Analyses and Data Handling | 4.0 |
| | | Conven | ntions | 13 |
| 6. | STLID | V D∩DI I | LATION ANALYSES | 1/ |
| 0. | 6.1. | | ew of Planned Study Population Analyses | |
| | 0.1. | Overvie | w of Flatified Study Fopulation Arialyses | 14 |
| 7. | SAFE | TY ANAL | YSES | 15 |
| | 7.1. | | e Events Analyses | |
| | 7.2. | | Laboratory Analyses | |
| 8. | | | INETIC ANALYSES | 16 |
| | 8.1. | | / Pharmacokinetic Analyses – Part A (Periods 1 – 3) and | |
| | | | (Periods 1 & 2) | |
| | | 8.1.1. | | |
| | | | 8.1.1.1. Drug Concentration Measures | |
| | | | 8.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 8.1.2. | Summary Measure | |
| | | 8.1.3. | Population of Interest | |
| | | 8.1.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.1.5. | Statistical Analyses / Methods | |
| | 0.0 | 0 | 8.1.5.1. Statistical Methodology Specification | 1/ |
| | 8.2. | | lary Pharmacokinetic Analyses - Part A (Periods 4-6), Part | 40 |
| | | 8.2.1. | Part C (Periods 3-6) | |
| | | 0.4.1. | Endpoint / Variables | |
| | | | 8.2.1.1. Drug Concentration Measures | |
| | | 8.2.2. | | |
| | | 8.2.3. | Summary Measure Population of Interest | |
| | | 8.2.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | ∪.∠.╅. | oratogy for intercurrent (i ost-ivandonization) Events | ∠∪ |


| 205017 |
|--------|
| 203017 |

| | | 8.2.5. | Statistical | Analyses / I | Methods | | | | 20 |
|---|---|---|---|---|---|---|---|---|---|
| | | | 8.2.5.1. | Statistical | Methodology | Specification | (Part | A) | 21 |
| | | | 8.2.5.2. | | | Specification | | | |
| | | | 8.2.5.3. | | | Specification | | | |
| | | | | | 0, | • | ` | , | |
| 9. | REFER | RENCES | | | | | | | 25 |
| 10. | APPEN | NDICES | | | | | | | 26 |
| | 10.1. | Appendix | 1: Protoco | ol Deviation | Managemen | t | | | 26 |
| | 10.2. | | | | | | | | |
| | | 10.2.1. | Protocol D | efined Sche | edule of Ever | nts | | | 27 |
| | 10.3. | Appendix | 3: Assess | ment Windo | ows | | | | 32 |
| | | | | | | s for Analyse | | | |
| | 10.4. | Appendix | 4: Study/T | reatment P | hases and A | dverse Events | s | | 33 |
| | | 10.4.1. | Treatment | Phases | | | | | 33 |
| | | 10.4.2. | Treatment | States | | | | | 33 |
| | | 10.4.3. | Treatment | States for A | AE Data | | | | 33 |
| | | 10.4.4. | Treatment | Phases for | Concomitan | t Medication | | | 33 |
| | 10.5. | Appendix | 5: Data Di | isplay Stand | dards & Hand | lling Conventi | ons | | 34 |
| | | 10.5.1. | | | | | | | |
| | | 10.5.2. | | | | | | | |
| | 10.6. | Appendix | 6: Derived | d and Trans | formed Data | | | | 36 |
| | | 10.6.1. | General | | | | | | 36 |
| | | 10.6.2. | Study Pop | ulation | | | | | 36 |
| | | 10.6.3. | Safety | | | | | | 37 |
| | | 10.6.4. | Pharmaco | kinetic | | | | | 37 |
| | | | 10.6.4.1. | Non-Comp | oartmental An | alysis | | | 37 |
| | 10.7. | Appendix | 7: Reporti | ng Standar | ds for Missing | g Ďata | | | 39 |
| | | 10.7.1. | | | | | | | |
| | | 10.7.2. | Handling of | of Missing D | )ata | | | | 39 |
| | | | 10.7.2.1. | Handling o | of Missing and | d Partial Date | s | | 39 |
| | 10.8. | Appendix | 8: Values | of Potential | Clinical Impo | ortance | | | 40 |
| | | 10.8.1. | Laboratory | / Values | | | | | 40 |
| | | 10.8.2. | ECG | | | | | | 41 |
| | | 10.8.3. | Vital Signs | 3 | | | | | 41 |
| | 10.9. | <b>Appendix</b> | 9: Pharma | acokinetic A | nalyses | | | | 42 |
| | | 10.9.1. | Systems | | | | | | 42 |
| | 10.10. | <b>Appendix</b> | 10: Abbre | viations & T | rade Marks. | | | | 43 |
| | 10.11. | | | | | | | | |
| | | 10.11.4. | | | | | | | |
| | | | | | | s Part A | | | |
| | | | | | | s Part B | | | |
| | | | | | | s Part C | | | |
| | | 10.11.5. | | | | | | | |
| | | | 10.11.5.1. | Safety Tab | oles Part A | | | | <u>5</u> 1 |
| | | | 10.11.5.3. | Safety Tab | oles Part C | | | | 57 |


| 10.11.6.1. Safety Figures | s Part A | 59 |
|---|---|---|
| 10.11.6.3. Safety Figures | Part C | 60 |
| Pharmacokinetic Tables | | 61 |
| 10.11.7.1. Pharmacokine | tic Tables Part A | 61 |
| 10.11.7.2. Pharmacokine | tic Tables Part B | 63 |
| 10.11.7.3. Pharmacokine | tic Tables Part C | 64 |
| Pharmacokinetic Figures | | 66 |
| 10.11.8.2. Pharmacokine | tic Figures Part B | 68 |
| ICH Listings | | 71 |
| 10.11.9.2. ICH Listings P | art B | 76 |
| 10.11.9.3. ICH Listing Pa | rt C | 82 |
| | 10.11.6.1. Safety Figures 10.11.6.2. Safety Figures 10.11.6.3. Safety Figures Pharmacokinetic Tables 10.11.7.1. Pharmacokine 10.11.7.2. Pharmacokine 10.11.7.3. Pharmacokine Pharmacokinetic Figures 10.11.8.1. Pharmacokine 10.11.8.2. Pharmacokine 10.11.8.3. Pharmacokine 10.11.8.3. Pharmacokine 10.11.9.1. ICH Listing Pa 10.11.9.1. ICH Listing Pa 10.11.9.3. ICH Listing Pa 10.11.9.3. ICH Listing Pa 10.11.10.1. Non-ICH Listings | 10.11.10.2. Non-ICH Listings Part B |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|----------------------|-------------|--------------|
| 2017N315344_00 | 07-Jul-2017 | Original |
| 2017N315344_01 | 18-Sep-2017 | Amendment 01 |
| 2017N315344_02 | 14-Jun-2018 | Amendment 02 |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 07-Jul-2017).

Protocol amendment 1: There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 18-Sep-2017).

Protocol amendment 2: Additional analyses were added for the inclusion of Part C that mirror what was specified for Part A (14-Jun-2018).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the single dose PK profile of GSK2982772 from each test minitab Modified Release (MR) formulation in a capsule (120 mg) compared to the IR formulation (120 mg) | GSK2982772 area under the curve from time zero to infinity (AUC(0-inf)), area under the curve from time zero to the last measurable concentration AUC(0-t), area under the curve from time zero to 24 hours AUC(0-24), area under the curve from time zero to 12 hours AUC(0-12), maximum observed concentration (Cmax), Concentration at 12 hours post-dose (C12h), Concentration at 24 hours post-dose (C24h) and ratio of Cmax: C12h and Cmax: C24h, relative bioavailability (Frelformulation) based on AUC and Cmax |
| To evaluate the single dose PK profile of GSK2982772 from a (matrix monolithic) MR tablet (240mg) compared to the IR formulation (240mg). | GSK2982772 AUC(0-inf), AUC(0-t), AUC(0-24),<br>AUC(0-12), Cmax, C12h, C24h, Cmax:C12h and<br>Cmax:C24h, Frel <sub>formulation</sub> based on AUC and Cmax. |
| Secondary Objectives | Secondary Endpoints |
| To assess the impact of high fat<br>meal on the PK of GSK2982772<br>following single dose | <ul> <li>GSK2982772 AUC(0-inf), AUC(0-t), Cmax, time to<br/>Cmax (Tmax), Frel<sub>FE</sub> based on AUC and Cmax,</li> </ul> |

| Objectives | Endpoints |
|---|---|
| administration of the selected minitab MR formulation in a capsule (120 mg) | • |
| To determine if there are any dose dependant changes in the absorption of GSK2982772 following repeat dose administration of the selected minitab MR formulation in a capsule at target daily doses of 30, 60 and 240 mg | <ul> <li>GSK2982772 AUC(0-24), Cmax, and Tmax if once daily (QD) dosing, on Day 1 and Day 3</li> <li>GSK2982772 AUC(0-12), AUC(12-24), Cmax, and Tmax after morning dose, Cmax and Tmax after evening dose if twice daily (BID) dosing, on Day 1 and Day 3</li> </ul> |
| To assess the impact of food on<br>the PK of GSK2982772 following<br>single dose administration of the<br>(matrix monolithic) MR tablet (dose<br>corrected, as appropriate). | <ul> <li>GSK2982772 AUC(0-inf), AUC(0-t) or AUC(0-24),<br/>Cmax, and time to Cmax (Tmax), Frel<sub>FE</sub> based on<br/>AUC and Cmax (dose corrected as appropriate).</li> </ul> |
| To determine if there are any dose dependent changes in the absorption of GSK2982772 following single dose administration or BID dose administration of the (matrix monolithic) MR tablet. | <ul> <li>GSK2982772 AUC(0-inf), AUC(0-t), AUC(0-24), Cmax, C24, Cmax:C24, and Tmax</li> <li>GSK2982772 AUC(0-12), C12, and Cmax:C12 if BID dosing</li> </ul> |
| To assess the safety and tolerability of single doses of GSK2982772 IR formulation and single and repeat doses of the (matrix monolithic) MR and minitab MR formulations in a capsule | <ul> <li>Adverse events (AEs)</li> <li>Clinical laboratory values (clinical chemistry, haematology and urinalysis)</li> <li>Vital sign measurements (blood pressure, heart rate, respiratory rate and body temperature)</li> <li>12-Lead electrocardiogram (ECG) monitoring</li> </ul> |
| Exploratory To assess the impact of a standard meal on the PK of GSK2982772 following administration of the selected minitab MR formulation in a capsule. | GSK2982772 AUC(0-inf), AUC(0-t), Cmax, Tmax, and Frel <sub>FE</sub> based on AUC and Cmax (dose corrected as appropriate). |

## 2.3. Study Design



| Overview of St | tudy Design and Key Features |
|---|---|
| | <ul> <li>(from Part A) following a 3 day repeat dosing of GSK2982772 at target daily doses of 30, 60 and 240mg (120mg, 240mg, 300mg actual daily doses).</li> <li>Part C – 6 period, sequential, 6-way fixed sequence design, with MR (matrix monolithic) formulations evaluated after single dose of GSK2982772 240mg in the fasted state.</li> </ul> |
| Dosing | Part A: |
| | <ul> <li>Single dose of GSK2982772 120mg will be evaluated. Periods 1, 2 and 3 will evaluate a slow minitab MR release duration, a fast minitab MR release formulation and IR tablet respectively. Periods 4, 5 and 6 will be flexible and depend on outcomes from Periods 1 to 3 and may be used to optimise the MR release durations and/or to evaluate the food effect.</li> <li>Part B:</li> </ul> |
| | <ul> <li>Target total daily doses of GSK2982772 30, 60 and 120mg QD or BID<br/>(depending on Part A findings) will be evaluated for 3 days. This<br/>corresponds to actual daily doses of 120, 240, and 300mg, respectively.<br/>Administration of the minitab MR formulation will either be in fasted state or<br/>with a standard meal (depending on Part A findings)</li> </ul> |
| | <ul> <li>Part C:</li> <li>Single dose of GSK2982772 240mg will be evaluated. Periods 1 and 2 will evaluate a (matrix monolithic) MR formulation and an IR tablet, respectively. Periods 3 through 6 will be flexible and the dosing regimen will be dependent on the outcome of Periods 1 and 2, and may evaluate higher doses, the impact of a high-fat meal, and/or standard meal after dosing or BID dosing.</li> </ul> |
| Time & Events | Refer to Appendix 2: Schedule of Activities |
| Treatment<br>Assignment | This is an open-label, non-randomised study. A treatment allocation list will take the place of the randomisation schedule, which will be developed by the sponsor using RandAll NG. |
| Interim<br>Analysis | <ul> <li>No formal interim analysis is planned for the study.</li> <li>Analysed PK data will be reviewed after completion of Periods 1 to 3 of part A which will guide Periods 4, 5 and 6.</li> <li>In Part C, there will be an interim review following completion of Periods 1 and 2 to determine the dose for Periods 3 and 4 (360 mg or 480 mg). Similarly, there will be an interim review following Periods 4 and 5 to determine dose, prandial state and and dosing regimen (QD or BID).</li> <li>Data will be reviewed following completion of Part A to determine the formulation, doses, dosing frequency (QD or BID) and prandial state for Part B.</li> </ul> |

# 2.4. Statistical Hypotheses / Statistical Analyses

No formal hypothesis will be tested. However, point estimates and corresponding 90% confidence intervals will be derived for the ratio between each minitab MR formulation relative to the IR formulation for the geometric mean of Cmax, Cmin, C12, C24, peak-to-trough ratio, AUC(0-inf), AUC(0-12), and AUC(0-24). PK parameters at the 12 hour time point will only be included if BID dosing is used.

### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal statistical analyses are planned.

#### Part A

After Periods 1 to 3 are complete, the PK and safety data will be analysed which will guide Periods 4, 5 and 6. Periods 4, 5 and 6 will be flexible and the dosing regimen will be dependent on the outcome of preceding periods. There will be the option to either optimise the MR release duration and/or to evaluate the impact of food on the selected MR minitab formulation in a capsule. There will also be the option to cancel Periods 5 and 6 if an optimal formulation is determined in Periods 1 or 2.

There will be an interim data review following final period of Part A to determine the formulation, doses, dosing frequency (QD or BID) and prandial state for Part B. The data, consisting of summary report of PK and safety endpoints will be sent to the sponsor by Quotient, from which the decision on formulation and prandial state selection or stopping the study will be made by the Quotient study team (i.e., PI, scientific lead and pharmacokineticist) and sponsor study team (as a minimum the sponsor's medical monitor, CPMS and GCSP). The decision will be documented and signed by the PI as per Quotient Clinical current SOP. Evidence of the decision will be retained in the ISF and GSK Trial Master File.

#### Part B

There will be no interim analysis during Part B of the study.

#### Part C

In Part C, there will be an interim review following completion of Periods 1 and 2 to determine the dose for Periods 3 and 4 (360 mg or 480 mg). Similarly, there will be an interim review following Periods 4 and 5 to determine dose, prandial state and dosing regimen (QD or BID). The data, consisting of summary report of PK and safety endpoints will be sent to the sponsor by Quotient, from which the decision on formulation and prandial state selection or stopping the study will be made by the Quotient study team (i.e., PI, scientific lead and pharmacokineticist) and sponsor study team (as a minimum the sponsor's medical monitor, CPMS and GCSP). The decision will be documented and signed by the PI as per Quotient Clinical current SOP. Evidence of the decision will be retained in the ISF and GSK Trial Master File.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects | All participants who were screened for eligibility and allocated a subject number. | Selected Study Population |
| Safety | All participants who receive at least 1 dose of study treatment and will be the population for reporting of safety and study population data. Participants will be analyzed according to the treatment they actually received. | Safety and Study Population |
| PK | Participants in the 'Safety Population' for whom a PK sample was obtained and analysed will be the population for reporting of PK data. | • PK |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP) 25-Sep-2018 Version 001. See Section 10.1 for further details.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Gr | oup Descriptions | |
|---|---|---|---|
| | RandAll NG | Data Displays for Re | eporting |
| Code | Description | Description | Order in TLF |
| Part A | | | |
| Α | GSK2982772 120mg minitab MR<br>RR1 oral single dose | MT-12h 120mg Fasted | 2 |
| В | GSK2982772 120mg minitab MR<br>RR2 oral single dose | MT-8h 120mg Fasted | 3 |
| С | GSK2982772 120mg IR oral single dose | IR 120mg Fasted | 1 |
| D | GSK2982772 120mg minitab MR<br>RR3 oral single dose | MT-12h 120mg Fed (Standard) | 4 |
| Е | GSK2982772 120mg minitab MR<br>RR4 oral single dose | n/a | 5 |
| F | GSK2982772 120mg minitab MR fed state | n/a | 6 |
| Part B | | | |
| G | GSK2982772 minitab MR Repeat<br>Dose 1 | MT-12h 120mg Fasted | 1 |
| Н | GSK2982772 minitab MR Repeat<br>Dose 2 | MT-12h 240mg Fasted | 2 |
| J | GSK2982772 minitab MR Repeat<br>Dose 3 | MT-12h 300mg Fed<br>(Standard) | 3 |
| Part C | | | |
| K | GSK2982772 240mg (matrix monolithic) MR oral single dose | MM-12h 240mg Fasted | 2 |
| L | GSK2982772 240mg IR oral single dose | IR 240mg Fasted | 1 |
| М | GSK2982772 360mg or 480mg<br>(matrix monolithic) MR oral single<br>dose | MM-12h 480mg Fasted | 3 |
| N* | GSK2982772 240mg (matrix monolithic) MR fed state | MM-12h 480mg Fed<br>(Standard) | 4 |
| Р | GSK2982772 360mg or 480mg<br>(matrix monolithic) MR delayed fed<br>(standard meal) or fed (high-fat<br>meal) | MM-12h 480mg Delayed<br>Fed (Standard) | 5 |
| Q | GSK2982772 dose tbd (matrix monolithic) MR QD or BID prandial state tbd. | MM-12h 240 mg Delayed<br>Fed (High-Fat) | 6 |

\* The randomization description for Period 4 of Part C (code N) indicates 240 mg, but the label has been updated to 480 mg to reflect the actual treatment administered.

### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Asses | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening Day -1 Day 1 (Pre-Dose) | | | |
| Safety | | | | |
| Vital signs | X | Χ | X | Day 1 (Pre-Dose) |
| 12-lead ECG | X | Χ | X | Day 1 (Pre-Dose) |
| Laboratory<br>(Haematology,<br>clinical chemistry<br>and urinalysis) | Х | Х | Х | Day 1 (Pre-Dose) |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 11: List of Data Displays.

In additional to GSK Core Data Standards, Lipids (Total Cholesterol and Triglycerides) outside the normal range will be summarised. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. Suicide risk monitoring including analyses of Colombia Suicide Severity Rating Scale (C-SSRS) and Possible Suicidality Related Adverse Event (PSRAE) will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays.

## 8. PHARMACOKINETIC ANALYSES

# 8.1. Primary Pharmacokinetic Analyses – Part A (Periods 1 – 3) and Part C (Periods 1 & 2)

## 8.1.1. Endpoint / Variables

### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.2 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin . All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Parts A and C F | Relative Bioavailability of MR vs IR |
| AUC <sub>(0-inf)</sub> | Area under the curve from time zero to infinity |
| AUC <sub>(0-t)</sub> 1 | Area under the curve from time zero to the last quantifiable concentration |
| AUC <sub>(0-24)</sub> | Area under the curve from time zero to 24 hours |
| AUC <sub>(0-12)</sub> [2] | Area under the curve from time zero to 12 hours, |
| AUC%extrap | Percentage of AUC extrapolated beyond the last measured time point. |
| t <sub>1/2</sub> | Terminal half-life |
| T <sub>lag</sub> | Time from dosing to first quantifiable concentration. |
| T <sub>max</sub> | Time of maximum observed concentration |
| C <sub>max</sub> | Maximum observed concentration |
| C <sub>24h</sub> | Concentration at 24 hours post-dose |
| C <sub>12h</sub> <sup>2</sup> | Concentration at 12 hours post-dose |
| C <sub>max</sub> :C <sub>12h</sub> <sup>2</sup> | Ratio of maximum and 12 hour concentrations |
| C <sub>max</sub> :C <sub>24h</sub> | Ratio of maximum and 24 hour concentrations |

#### NOTES:

- Additional parameters may be included as required.
- No log transformation for Tmax nor any ratio (relative) endpoint.
- [1]: AUC<sub>(0-t)</sub> if AUC<sub>(0-inf)</sub> cannot be derived
- [2]: If BID

## 8.1.2. Summary Measure

For each release rate in Periods 1 through 3 of Part A, and Periods 1 and 2 of Part C, descriptive statistics (n, arithmetic mean, standard deviation [SD], 95% CI, minimum, median and maximum,) will be calculated by treatment for all PK concentrations over

time and for the derived PK parameters. In addition, for loge-transformed PK parameter variables geometric mean, 95% CI, and %CV<sub>b</sub> will be provided, where %CV<sub>b</sub> =(100 \*  $\sqrt{\exp(SD2)}$  -1)) and SD is the standard deviation of log-transformed data.

#### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

- Participant study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.
- Withdrawn participants may be replaced in the study. Replacement participants enrolled will be dosed with the next planned treatment of the withdrawn participant, and they will not receive any treatment that the withdrawn participant has already received with the exception of the need to increase participant numbers to obtain the minimum number of evaluable participants required for interim decisions, and to obtain data in any other treatment that is required for a valid comparison. Replacement participants will receive the required treatments in the same order as planned for the original participant and the minimum washout period will be respected with regard to the timing of dosing of the IR formulation.
- All available data from participants who were withdrawn from the study will be listed
  and all available planned data will be included in summary tables and figures, unless
  otherwise specified.

### 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### **Endpoint (log scale)**

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub> if AUC<sub>(0-inf)</sub> cannot be derived
- AUC<sub>(0-12)</sub> if BID
- AUC<sub>(0-24h)</sub>

- C<sub>max</sub>
- C<sub>12h</sub> if BID
- C<sub>24h</sub>

#### **Model Specification**

- For each endpoint a mixed model will be fit with 3 observations per participant expected in Part
  A, and 2 observations per participant in Part C. The model will contain formulation as a fixed,
  categorical effect, and a random intercept for subject.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

## **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data
- In the event the model fails to converge, the RANDOM statement will be removed and alternative covariance structures such as CS, CSH, or UN for the R matrix will be used by specifying 'type=' on the REPEATED line. Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.
- If outliers are detected, an additional table will be produced with outlying observations omitted.

#### **Model Results Presentation**

- Point estimates and corresponding 90% CI will be computed for the differences in the endpoint for each GSK2982772 MR formulation vs GSK2982772 IR formulation.
- The relative bioavailability ratio, Frel<sub>formulation</sub>, and 90% CI will be calculated by back-transforming the difference between the least square means for each of the two formulation comparisons. See Section 10.6.4

# 8.2. Secondary Pharmacokinetic Analyses - Part A (Periods 4-6), Part B, and Part C (Periods 3-6)

#### 8.2.1. Endpoint / Variables

#### 8.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.2 Reporting Standards for Pharmacokinetic)

#### 8.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Part A - Food | Effect |
| AUC <sub>(0-inf)</sub> | Area under the curve from time zero to infinity |
| $AUC_{(0-t)}^{1}$ | Area under the curve from time zero to last quantifiable concentration |
| AUC <sub>(0-12)</sub> <sup>2</sup> | Area under the curve from time zero to 12 hours |
| AUC <sub>(0-24)</sub> 3 | Area under the curve from time zero to 24 hours |
| $C_{max}$ | Maximum observed concentration |
| $C_{12h}^2$ | Concentration at 12 hours post-dose |
| C <sub>24h</sub> | Concentration at 24 hours post-dose |
| $C_{\text{max}} : C_{12h}{}^2$ | Ratio of maximum and 12 hour concentrations |
| C <sub>max</sub> :C <sub>24h</sub> | Ratio of maximum and 24 hour concentrations |
| T <sub>max</sub> | Time of maximum observed concentration |
| Part B – Repe | eat Dose |
| AUC <sub>(0-12)</sub> <sup>2</sup> | Area under the curve from time zero to 12 hours |
| AUC <sub>(12-24)</sub> <sup>2</sup> | Area under the curve from time 12hours to 24 hours |
| AUC <sub>(0-24)</sub> 3 | Area under the curve from time zero to 24 hours |
| C <sub>max</sub> | Maximum observed concentration |
| $C_{12h}^2$ | Concentration at 12 hours post-dose |
| C <sub>24h</sub> | Concentration at 24 hours post-dose |
| $C_{\text{max}} : C_{12h}{}^2$ | Ratio of maximum and 12 hour concentrations |
| C <sub>max</sub> :C <sub>24h</sub> | Ratio of maximum and 24 hour concentrations |
| T <sub>max</sub> | Time of maximum observed concentration |
| Part C - High | Dose Food Effect |
| AUC <sub>(0-inf)</sub> | Area under the curve from time zero to infinity |
| $AUC_{(0-t)}^{1}$ | Area under the curve from time zero to the last quantifiable concentration |
| AUC <sub>(0-24)</sub> 3 | Area under the curve from time zero to 24 hours |
| AUC <sub>(0-12)</sub> 1 | Area under the curve from time zero to 12 hours |
| T <sub>max</sub> | Time of maximum observed concentration |
| C <sub>max</sub> | Maximum observed concentration |
| C <sub>min</sub> | Minimum observed concentration |
| C <sub>24h</sub> | Concentration at 24 hours post-dose |
| C <sub>12h</sub> <sup>2</sup> | Concentration at 12 hours post-dose |

| Parameter | Parameter Description |
|---|---|
| $C_{\text{max}}:C_{12h}^2$ | Ratio of maximum and 12 hour concentrations |
| C <sub>max</sub> :C <sub>24h</sub> | Ratio of maximum and 24 hour concentrations |

#### NOTES:

- Additional parameters may be included as required.
- No log transformation for Tmax nor any ratio (relative) endpoint.
- [1]: AUC<sub>(0-t)</sub> if AUC<sub>(0-inf)</sub> cannot be derived
- [2]: If BID formulation.
- [3]: QD formulation only.

#### 8.2.2. Summary Measure

For each fed/fasted state in Parts A and C, and for day 1 and day 3 of every dose (period) in Part B, descriptive statistics (n, arithmetic mean, standard deviation [SD], 95% CI, minimum, median and maximum,) will be calculated by treatment for all PK concentrations over time and for the derived PK parameters. In addition, for loge-transformed PK parameter variables geometric mean, 95% CI and %CV<sub>b</sub> will be provided, where %CV<sub>b</sub> =(100 \*  $\sqrt{\text{(exp(SD2) -1)}}$ ) and SD is the standard deviation of log-transformed data.

For Part B, log-scale dose normalized  $C_{max}$ ,  $C_{12h \text{ (for BID)}}$ ,  $C_{24h}$ ,  $AUC_{(0-12)}$  (for BID dosing) AUC(12-24) (for BID dosing), and  $AUC_{(0-24)}$  will also be summarized. Plots of dose vs log-scale dose normalised  $AUC_{(0-24)}$ ,  $(AUC_{(0-12)}$  and  $AUC_{(12-24)}$  for BID dosing),  $C_{12h \text{ (for BID)}}$ ,  $C_{24h}$ , and  $C_{max}$  (after morning and evening doses if BID dosing) will be generated to determine if there are any dose dependent changes in the absorption of GSK2982772 following repeat dose administration of the selected minitab MR formulation.

#### 8.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

• See Section 8.1.4.

## 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.2.5.1. Statistical Methodology Specification (Part A)

#### **Endpoint (log scale)**

- AUC<sub>(0-inf)</sub>
- AUC<sub>(0-t)</sub> if AUC<sub>(0-inf)</sub> cannot be derived
- Cmax

#### **Model Specification**

- For each endpoint a mixed model will be fit with 2 observations per subject expected. The
  model will contain state [[fed/fasted] as a fixed, categorical effect and a random intercept for
  subject.
- The Kenward & Roger (KR) degreed of freedom approach will be used.

## **Model Checking & Diagnostics**

See Section 8.1.5.1

### **Model Results Presentation**

- Point estimates and corresponding 90% CI will be computed for the differences in the endpoint for GSK2982772 MR formulation (120 mg) taken in the fed state (test) vs in the fasted state (reference) using the residual error from the model (MSE).
- The point and interval estimates on the log-scale will then be exponentially back transformed to give estimates of the ratios of geometric means, Frel<sub>FE</sub>, and 90% CI. See Section 10.6.4

#### **Endpoint**

Tmax

#### **Model Specification**

- Exact non-parametric Hodges-Lehmann estimation of location shift will be fitted.
- Only the dose of GSK2982772 administered under both fed and fasted conditions will be used.

#### **Model Results Presentation**

- GSK2982772 MR formulation in fed (test) will be compared to fasted (reference) state.
- Median difference and 90% CI for median difference will be presented.

#### 8.2.5.2. Statistical Methodology Specification (Part B)

#### **Endpoint (log scale)**

- AUC<sub>(0-24h)</sub> (QD)
- AUC<sub>(0-12h)</sub> (if BID)
- AUC<sub>(12-24h)</sub> (if BID)
- Cmax (morning) (QD or BID)
- Cmax (evening) (if BID)

#### **Model Specification**

- For each endpoint a mixed model will be fit with 6 observations per subject expected. The
  model will contain dose (120, 240, 300) and day (1,3) as fixed, categorical effects, and their
  interaction.
- A direct product (UN@CS) covariance pattern will be fit using period and day (in that order) as the effects in the REPEATED statement.
- The Kenward & Roger (KR) degrees of freedom approach will be used.

#### **Model Checking & Diagnostics**

- See Section 8.1.5.1. Additionally, in the event the model fails to converge a compound symmetric covariance pattern will be fit using day\*dose as the effect on the REPEATED statement, with type=CS, group=period, and subject id specified in the subject= option to account for the correlation between days within period. A random intercept effect will also be included to account for the correlation between days across period.
- In the event the above model fails to converge, a compound symmetric covariance pattern will be fit using day\*dose as the effect on the REPEATED statement, with type=CS and subject id specified in the subject= option. A random period effect will also be included.
- In the event the above model fails to converge, a compound symmetric covariance pattern will be fit using day\*dose as the effect on the REPEATED statement, with type=CS and subject id specified in the subject= option.
- In the event the above model fails to converge, all other covariance patterns will be explored, including unstructured.
- If outliers are detected, an additional table will be produced with outlying observations omitted.

### **Model Results Presentation**

- Point estimates and corresponding 90% CI will be computed for the differences in the endpoint between Day 1 and Day 3 for Period 1 (120mg daily), Period 2 (240mg daily), and Period 3 (300mg daily) for GSK2982772 minitab MR dose.
- The point and interval estimates on the log-scale will then be exponentially back transformed to give estimates of the ratios of geometric means, Frel<sub>Dav</sub>, and 90% Cl. See Section 10.6.4

#### 8.2.5.3. Statistical Methodology Specification (Part C)

Bioavailability of Food Effect

### **Endpoint (log scale)**

- AUC(0-inf)
- AUC(0-t) if AUC(0-inf) not available
- Cmax
- •

### **Model Specification**

 For each endpoint a mixed model will be fit with 5 observations per subject expected. The model will contain dose (240mg, 480mg) and prandial state [fed (standard)/delayed fed

- (standard)/delayed fed (high-fat)/fasted] as a fixed, categorical effect and a random intercept for subject.
- A direct product (UN@CS) covariance pattern will be fit using dose and state (in that order) as the effects in the REPEATED statement.
- The Kenward & Roger (KR) degrees of freedom approach will be used.

#### **Model Checking & Diagnostics**

• See Section 8.1.5.1.

#### **Model Results Presentation**

- Point estimates and corresponding 90% CI will be computed for the differences in the endpoint for GSK2982772 MR formulation (240 mg or 480 mg) taken in the fed state (test) vs in the fasted state (reference) using the residual error from the model (MSE).
- The point and interval estimates on the log-scale will then be exponentially back transformed to give estimates of the ratios of geometric means, Frel<sub>FE</sub>, and 90% Cl. See Section 10.6.4

#### **Endpoint**

Tmax

#### **Model Specification**

- Exact non-parametric Hodges-Lehmann estimation of location shift will be fitted.
- Only the dose of GSK2982772 administered under both fed and fasted conditions will be used.

#### **Model Results Presentation**

- GSK2982772 MR formulation in fed (test) state will be compared to fasted (reference) state.
- Median difference and 90% CI for median difference will be presented.

#### Bioavailability of Dose

#### **Endpoint (log scale)**

- AUC(0-inf)
- AUC(0-t) if AUC(0-inf) not available
- AUC(0-24)
- Cmax
- C24

#### **Model Specification**

- For each endpoint a mixed model will be fit with 2 observations per subject expected. The
  model will contain dose (480 mg and 240 mg in the fasted state) as a fixed, categorical effect,
  and a random intercept for subject.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

# **Model Checking & Diagnostics**

See Section 8.1.5.1.

#### **Model Results Presentation**

- Point estimates and corresponding 90% CI will be computed for the differences in the endpoint for GSK2982772 MR dose (480 mg vs 240 mg) using the residual error from the model (MSE).
- The point and interval estimates on the log-scale will then be exponentially back transformed to give estimates of the ratios of geometric means, Frel<sub>DOSE</sub>, and 90% CI. See Section 10.6.4

#### **Endpoint**

Tmax

#### **Model Specification**

- Exact non-parametric Hodges-Lehmann estimation of location shift will be fitted.
- Only GSK2982772 administered at 240 mg and 480 mg.

#### **Model Results Presentation**

- GSK2982772 MR formulation at 480 mg (test) state will be compared to 240 mg (reference).
- Median difference and 90% CI for median difference will be presented.

## 9. REFERENCES

GlaxoSmithKline Document Number 2017N315344\_02. A three part, non-randomised, open label study designed to assess the pharmacokinetics of GSK2982772 following administration of minitab modified release formulations in a capsule relative to an immediate release reference tablet formulation (Part A), the pharmacokinetics of escalating, repeat doses of a selected minitab modified release prototype (Part B), and the pharmacokinetics of GSK2982772 following administration of modified release tablet formulations in the fed and fasted state (Part C) in healthy participants. Effective Date: 14-JUN-2018

Hauschke D1, Steinijans VW, Diletti E. A distribution-free procedure for the statistical analysis of bioequivalence studies. *Int J Clin Pharmacol Ther Toxicol*, 1990;28(2):72-8.

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

Schedule of Activities for Parts A and C

| Procedure | Screening<br>(up to 28 days before Day 1) | Treatme | nt Period 1, 2,<br>Day | 3, 4, 5, 6 | Follow-up/Study<br>Discontinuation<br>(7 days post last dose) | Notes |
|---|---|---|---|---|---|---|
| | | -1 | 1 | 2 | | |
| Informed consent | X | | | | | |
| Inclusion and exclusion criteria <sup>1</sup> | Х | | | | | <ol> <li>Recheck clinical status<br/>before 1st dose of study<br/>medication.</li> </ol> |
| Demography | X | | | | | |
| Demonstrate ability to swallow size 0-00 capsules | Х | | | | | |
| Full physical examination including height and weight | Х | | | | | |
| Brief physical examination | | х | | X2 | Х | Discharge (32 h post-dose for Treatment Period 1, 2, 4, 5 and 6 in Part A and Treatment Period 1, 3, 4, 5 and 6 in Part C 24 h post-dose for Treatment Period 3 in Part A and Treatment Period 2 Part C) |
| Medical history (includes substance usage) <sup>3</sup> | Х | | | | | <ol> <li>Substances: Drugs,<br/>Alcohol, tobacco and<br/>caffeine</li> </ol> |
| Past and current medical conditions | Х | | | | | |


### 205017

| Procedure | Screening<br>(up to 28 days before Day 1) | Treatme | ent Period 1, 2,<br>Day | 3, 4, 5, 6 | Follow-up/Study<br>Discontinuation<br>(7 days post last dose) | Notesa |
|---|---|---|---|---|---|---|
| | ., | -1 | 1 | 2 | | |
| Follide Stimulating Hormone (FSH) (as needed in women of non-childbearing potential only) | Х | | | | | |
| Serum pregnancy test (WOCBP only) | X | | | | X | |
| Urine pregnancy test (WOCBP only) | | х | | | | |
| Human Immunodefeciency Virus (HIV),<br>Hepatitis B and C screening <sup>4</sup> | х | | | | | If test otherwise<br>performed within 3<br>months prior to first dose<br>of study treatment, testing<br>at screening is not<br>required |
| Tuberculosis (TB) Test | X | | | | | |
| Urine drug screen | Х | X | | | | |
| Alcohol breath test | Х | х | | | | |
| Carbon monoxide breath test | Х | Х | | | | |
| Laboratory assessments (haematology, dinical chemistry and urinalysis) | Х | Х | X <sup>5</sup> | X5 | х | Pre-dose (Treatment<br>Period 1 only) and 24 h<br>post-dose<br>Allowable windows in<br>Section 9.4.4 |
| Glomerular filtration rate | X | | | | | |
| C-reactive protein (CRP) | Х | | | | | |

| Procedure | Screening<br>(up to 28 days before Day 1) | Treatme | ent Period 1, 2,<br>Day | 3, 4, 5, 6 | Follow-up/Study<br>Discontinuation<br>(7 days post last dose) | Notes <sup>a</sup> |
|---|---|---|---|---|---|---|
| | | -1 | 1 | 2 | | |
| 12-lead ECG | Χę | Х | X <sup>7</sup> | X8 | х | In triplicate Pre-dose and 2 and 12 h post-dose 24 h post-dose Allowable windows in Section 9.4.3 |
| Vital signs | Х | Х | Xa | X <sup>10</sup> | Х | Pre-dose and 2 and 12 h post-dose 10. 24 h post-dose Allowable windows in Section 9.4.2 |
| Study treatment | | | X | | | |
| AE review | | <b>←=====</b> | | | X | |
| Serious AE (SAE) review | X | <b>←</b> | | | X | |
| Concomitant medication review | | <b>←</b> | | Х | | |
| PK blood sample collection | | | X11 | X11 | | 11. Time points in Table 2 |

<sup>&</sup>lt;sup>a</sup> The timing of assessments may be amended in Part C if BID dosing is selected for any of the regimens.

# Pharmacokinetic Blood Sample Collection Times for Parts A and C

| | Part A Treatment Periods 1, 2, 4, 5 and 6 (MR Formulations) Part C Treatment Periods 1, 3, 4, 5 and 6 (MR Formulations) | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time (h) | Pre-<br>dose | 0 | 2 | 4 | 6 | 8 | 10 12 | 14 | 16 | 18 | 20 | 22 24 | 2 | 26 | 28 3 | 0 | 32 |
| Dosing | | Χ | | | | | | | | | | | | | | | |
| PK sampling | Χ | | Χ | Χ | X | Χ | X X | X | X | Χ | X | ( X | Х | ( | X ) | ( | X |
| | Part A: Treatment Period 3 (IR Formulation) Part C: Treatment Period 2 (IR Formulation) | | | | | | | | | | | | | | | | |
| Time (h) | Pre-<br>dose | 0 | 0.33 | 0. | .66 | 1 | 1.5 | 2 | 3 | 4 | 6 | 8 | 10 | | 12 | 24 | |
| Dosing | | Χ | | | | | | | | | | | | | | | |
| PK sampling | X | | Χ | X | | X | X | Χ | Χ | Χ | X | X | X | | Χ | X | |

<sup>&</sup>lt;sup>a</sup> PK sampling schedule may be amended in Part C if BID dosing is selected for any of the regimens. If BID dosing is employed the number of PK samples may be reduced i.e. some of the samples between 14 and 24 h may not be required. In addition, the 12 h sample will be taken prior to administering the second daily dose.

# Schedule of Activities for Part B

| Procedure | Screening<br>(up to 28 days before Day 1) | Treatment Period 1, 2, 3<br>Day | | | | | Follow-up/Study<br>Discontinuation<br>(7 days post last<br>dose) | | Notes |
|---|---|---|---|---|---|---|---|---|---|
| | | -1 | 1 | 2 | 3 | 4 | | | |
| Informed consent | X | | | | | | | | |
| Inclusion and exclusion criteria¹ | Х | | | | | | | 1. | Recheck clinical status before<br>1st dose of study medication. |
| Demography | х | | | | | | | | |
| Demonstrate ability to swallow size 0-00 capsules | Х | | | | | | | | |
| Full physical examination including height and weight | Х | | | | | | | | |
| Brief physical examination | | Х | | | | X2 | х | 2. | Discharge (24 h after the last dose) |
| Medical history (includes substance usage) <sup>3</sup> | Х | | | | | | | 3. | Substances: Drugs, Alcohol, tobacco and caffeine |
| Past and current medical conditions | Х | | | | | | | | |
| FSH (as needed in women of non-<br>childbearing potential only) | Х | | | | | | | | |
| Serum pregnancy test (WOCBP only) | Х | | | | | | Х | | |
| Urine pregnancy test (WOCBP only) | | Х | | | | | | | |


### 

| Procedure | Screening<br>(up to 28 days before Day 1) | | Treatme | ent Perio<br>Day | d 1, 2, 3 | | Follow-up/Study<br>Discontinuation<br>(7 days post last<br>dose) | Notes | |
|---|---|---|---|---|---|---|---|---|---|
| HIV, Hepatitis B and C screening <sup>4</sup> | X | -1 | 1 | 2 | 3 | 4 | | 4. | If test otherwise performed<br>within 3 months prior to first<br>dose of study treatment,<br>testing at screening is not<br>required |
| Tuberculosis Test | X | | | | | | | | |
| Urine drug screen | Х | X | | | | | | | |
| Alcohol breath test | X | Х | | | | | | | |
| Carbon monoxide breath test | X | Х | | | | | | | |
| Laboratory assessments (haematology, clinical chemistry and urinalysis) | x | x | X <sup>5</sup> | | | X <sup>6</sup> | х | 5.<br>6. | Pre-dose<br>24 h after the last dose<br>Allowable windows in Section<br>9.4.4 |
| Glomerular filtration rate | х | | | | | | | | |
| CRP | х | | | | | | | | |
| ANA | х | | | | | <b>X</b> <sup>7</sup> | | 7. | 24 h after the last dose |
| 12-lead ECG | Χs | x | X <sub>9</sub> | X <sup>10</sup> | X9 | X <sup>11</sup> | х | 10. | In triplicate Pre-dose and 2 and 12 h post-dose Pre-dose 24 h after the last dose Allowable windows in Section 9.4.3 Time points may be subject to change depending on results from Part A |
| Vital signs | X | Х | X <sup>12</sup> | X <sup>13</sup> | X <sup>12</sup> | X14 | х | 13.<br>14. | Pre-dose and 2 and 12 h post-dose Pre-dose 24 h after the last dose Allowable windows in Section 9.4.2 Time points may be subject to change depending on results from Part A |
| Columbia Suicide Risk questionnaire | Х | | X15 | | | X <sup>16</sup> | | | Pre-dose<br>24 h after last dose of each<br>period |
| Study treatment | | | X | Х | X | | | | |
| AE review | | <del></del> | | | | <del>&gt;</del> | Х | | |
| SAE review | х | <del></del> | | | | <del>&gt;</del> | Х | | |
| Concomitant medication review | | ← | | | <del>&gt;</del> | Х | | | |
| PK blood sample collection | | | X17 | X17 | X17 | X <sup>17</sup> | | 17. | Time points in Table 4 |

#### Pharmacokinetic Blood Sample Collection Times for Part B

| | | Periods 1, 2 and 3 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Days 1 and 3 | | | | | | | | | | | | |
| Time (h) | Pre-<br>dose | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 |
| Dosinga | | X | | | | | | | | | | | | |
| PK sampling <sup>b</sup> | X | | Χ | X | Χ | Χ | Χ | X | Χ | Χ | Χ | X | Χ | Χc |

<sup>&</sup>lt;sup>a</sup> Subjects will be dosed on Days 1, 2 and 3; however, no PK samples will be taken post-dose on Day 2

PK samples should take priority over other procedures scheduled at the same time point. As guidance, the preferred order of assessments is:



Electrocardiograms (ECGs) should be taken prior to vital signs when both measurements are scheduled at the same time point. Other assessments, e.g. physical examinations etc, will be performed within the required time windows. All safety assessments will be timed and performed relative to the start of dosing.

<sup>&</sup>lt;sup>b</sup> PK sampling schedule may be amended based upon the PK data from Part A and/or if BID dosing is selected for Part B. If BID dosing is employed the number of PK samples may be reduced i.e. some of the samples between 14 and 24 h may not be required. In addition, the 12 h sample will be taken prior to administering the second daily dose.

<sup>&</sup>lt;sup>c</sup> Day 1 24 h post-dose sample should be taken prior to dosing on Day 2.

# 10.3. Appendix 3: Assessment Windows

# 10.3.1. Definitions of Assessment Windows for Analyses

No Assessment Windows will be defined for Analysis, and summaries and analyses will be based on nominal visits.

# 10.4. Appendix 4: Study/Treatment Phases and Adverse Events

#### 10.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to dosing.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date <sup>[1]</sup> ≤ Study Treatment Start Date <sup>[1]</sup> |
| On-Treatment | Study Treatment Start Date <sup>[1]</sup> < Date <sup>[1]</sup> ≤ Study Treatment Stop Date <sup>[1]</sup> |
| Post-Treatment | Date <sup>[1]</sup> > Study Treatment Stop Date <sup>[1]</sup> |

<sup>[1]</sup> Datetime if Time is present for assessments or events

#### 10.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 10.4.3. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

## 10.4.4. Treatment Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

## 10.5.1. Reporting Process

| Software | |
|---|---|
| The currently su | The currently supported versions of SAS software and WIN-NonLin will be used. |
| Reporting Area | Reporting Area |
| HARP Server | : UK1SALX00175 |
| HARP Area | Final |
| | : \arprod\gsk2982772\ mid205017\final_01 |
| QC Spreadsheet | : \arwork\gsk2982772\mid205017\documents |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated for SAC tables. | |

### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### **Formats**

- All data will be reported according to the actual treatment the subject receives unless otherwise states.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
- PK Summary Statistics: 3 significant figures for the lowest value of each PK parameter. The summary statistics for higher values will be reported to the same number of decimal places as the lowest value

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.

- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- If there are two values within a time window (as per Section 10.3.1) the value closest to the target day
  for that window will be used. If values are the same distance from the target, then the mean will be
  taken.
- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 10.6.2. Study Population

## **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

## **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.
## 10.6.3. Safety

### **ECG Parameter**

### **RR** Interval

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{\dot{Q}T}{\sqrt{\frac{RR}{1000}}} \qquad QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places= '< x ' becomes x 0.01
  - Example 2: 1 Decimal Places = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Places = '< x' becomes x 1</p>

### 10.6.4. Pharmacokinetic

## 10.6.4.1. Non-Compartmental Analysis

The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices using WinNonlin Version 6.3 or higher.

## **Pharmacokinetic Endpoints**

## AUC(0-t)

Area under the concentration-time curve from time zero to the time of the last quantifiable concentration
(C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log
trapezoidal rule for each decremental trapezoid.

## **Pharmacokinetic Endpoints**

## AUC(0-∞) (Day 1)

• Area under the concentration-time curve extrapolated to infinity will be calculated as:

$$AUC = AUC(0-t) + C(t) / lambda_z$$

where lambda z is the terminal phase rate constant.

## AUC(0-24) for QD dosing

Area under the concentration-time curve from time zero to 24 h post dose will be calculated using the linear trapezoidal rule for each incremental trapezoid.

## AUC(0-12) for BID dosing

Area under the concentration-time curve from time zero to 12 h post dose will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.

## AUC(12-24) for BID dosing

Area under the concentration-time curve from time 12 h to 24 h post dose will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.

### **AUC%extrap**

Percentage of AUC extrapolated beyond the last measured time point

### $C_{\text{max}}$

Maximum observed concentration, determined directly from the concentration-time data

### C<sub>12h</sub> for BID dosing

Observed concentration at 12 hours, determined directly from the concentration-time data

### C<sub>24h</sub>

Observed concentration at 24 hours, determined directly from the concentration-time data

### Tmax

Time to reach Cmax, determined directly from the concentration-time data.

## Tlag

Time from dosing at which GSK2982772 was first quantifiable in a concentration vs time profile

### t1/2

Terminal half-life

### **Notes**

Additional parameters may be included as required

## Relative Bioavailability (Frel)

• Frel will be calculated as follows:

$$Frel = \frac{GeoMean\{AUC\ or\ C_{max}(test)\}}{GeoMean\{AUC\ or\ C_{max}(reference)\}} \times 100$$

Frel will be calculated using  $AUC_{(0-inf)}$  and  $C_{max}$ . If for any reason the  $AUC_{(0-inf)}$  is not calculable then an alternative AUC such as  $AUC_{(0-last)}$ ,  $AUC_{(0-\mathbb{T})}$  or AUC over a partial area may be used. The following comparisons will be made:

- MR Formulation (test) vs IR Formulation (reference)
- Fed (test) vs Fasted (reference)
- Day 3 vs Day 1 (reference)

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as one who completes all phases of the study including the last scheduled procedure shown in the SoA i.e. the follow-up visit. |
| | Withdrawn subjects may be replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| White Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | | | 1.3 X ULN |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5x ULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 10.8.2. ECG

| ECG Parameter | Units | Clinical Co | Clinical Concern Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| | | ≤ 450 | |
| Absolute QTc Interval | msec | > 450 | <480 |
| ADSOIDLE QTC IIILEIVAI | | ≥ 480 | <500 |
| | | ≥ 500 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | Change from Baseline | | |
| | msec | ≤ 30 | |
| Increase from Baseline QTc | msec | > 30 | <60f |
| | msec | ≥ 60 | |

# 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

- 10.9. Appendix 9: Pharmacokinetic Analyses
- 10.9.1. Systems

N/A

# 10.10. Appendix 10: Abbreviations & Trade Marks

# 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Friderica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 10.10.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

None

# Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

## 10.11. Appendix 11: List of Data Displays

## 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables Figures | |
|------------------|-----------------------|------------|
| Study Population | 1.1 to 1.n 1.1 to 1.n | |
| Safety | 2.1 to 2.n | 2.1 to 2.n |
| Pharmacokinetic | 3.1 to 3.n | 3.1 to 3.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

## 10.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 10.11.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

## NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.11.4. Study Population Tables

## 10.11.4.1. Study Population Tables Part A

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of Subject Disposition: Part A | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.2. | All Subjects | ES6 | Summary of Reasons for Screen Failure: Part A | Journal Requirements | SAC |
| Protoc | ol Deviation | | | | |
| 1.3. | Safety | DV1 | Summary of Important Protocol Deviations: Part A | ICH E3 | SAC |
| 1.4. | All Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Deviations: Part A | IDSL | SAC |
| Popula | tion Analysed | | | | |
| 1.5. | All Subjects | SP1 | Summary of Study Populations and Exclusions: Part A | IDSL | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.34. | All Subjects | DM11 | Summary of Age Ranges: Part A | ICH E3, GSK CTR, FDAAA, EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years'). | SAC |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics: Part A | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.7. | Safety | DM5 | Summary of Race and Racial Combinations: Part A | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | SAC |
| 1.8. | Safety | DM6 | Summary of Race and Racial Combination Details: Part A | ICH E3, FDA | SAC |

| Study F | Population Tab | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.9. | Safety | MH4 | Summary of Current/Past Medical Conditions: Part A | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.10. | Safety | CM1 | Summary of Concomitant Medications: Part A | ICH E3 | SAC |
| Exposu | ire and Treatmo | ent Compliance | | | |
| 1.11. | Safety | EX1 | Summary of Exposure to Study Treatment: Part A | ICH E3 Dose and/or time on treatment, as applicable. | SAC |

# 10.11.4.2. Study Population Tables Part B

| Study Popu | lation Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject Dis | position | | | | |
| 1.12. | Safety | ES1A | Summary of Subject Disposition: Part B | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.13. | All Subjects | ES6 | Summary of Reasons for Screen Failure: Part B | Journal Requirements | SAC |
| Protocol De | eviation | | | | |
| 1.14. | Safety | DV1 | Summary of Important Protocol Deviations: Part B | ICH E3 | SAC |
| 1.15. | All Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Deviations: Part B | IDSL | SAC |
| Population | Analysed | | | | |
| 1.16. | All Subjects | SP1 | Summary of Study Populations and Exclusions: Part B | IDSL | SAC |
| Demograph | nic and Baselin | e Characteris | tics | | |
| 1.35. | All Subjects | DM11 | Summary of Age Ranges: Part B | ICH E3, GSK CTR, FDAAA, EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years'). | SAC |
| 1.17. | Safety | DM1 | Summary of Demographic Characteristics: Part B | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.18. | Safety | DM5 | Summary of Race and Racial Combinations: Part B | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | SAC |
| 1.19. | Safety | DM6 | Summary of Race and Racial Combination Details: Part B | ICH E3, FDA | SAC |

| Study Popul | ation Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior and Co | ncomitant Me | dications | | | |
| 1.20. | Safety | MH4 | Summary of Current/Past Medical Conditions: Part B | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.21. | Safety | CM1 | Summary of Concomitant Medications: Part B | ICH E3 | SAC |
| Exposure ar | d Treatment C | ompliance | | | |
| 1.22. | Safety | EX1 | Summary of Exposure to Study Treatment: Part B | ICH E3 Dose and/or time on treatment, as applicable. | SAC |

# 10.11.4.3. Study Population Tables Part C

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.23. | Safety | ES1A | Summary of Subject Disposition: Part C | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.24. | All Subjects | ES6 | Summary of Reasons for Screen Failure: Part C | Journal Requirements | SAC |
| Protoc | ol Deviation | | | | |
| 1.25. | Safety | DV1 | Summary of Important Protocol Deviations: Part C | ICH E3 | SAC |
| 1.26. | All Subjects | IE2 | Summary of Inclusion/Exclusion Criteria Deviations: Part C | IDSL | SAC |
| Popula | tion Analysed | | | | |
| 1.27. | All Subjects | SP1 | Summary of Study Populations and Exclusions: Part C | IDSL | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.36. | All Subjects | DM11 | Summary of Age Ranges: Part C | ICH E3, GSK CTR, FDAAA, EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years'). | SAC |
| 1.28. | Safety | DM1 | Summary of Demographic Characteristics: Part C | ICH E3, GSK CTR, FDAAA, EudraCT | SAC |
| 1.29. | Safety | DM5 | Summary of Race and Racial Combinations: Part C | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | SAC |
| 1.30. | Safety | DM6 | Summary of Race and Racial Combination Details: Part C | ICH E3, FDA | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 1.31. | Safety | MH4 | Summary of Current/Past Medical Conditions: Part C | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.32. | Safety | CM1 | Summary of Concomitant Medications: Part C | ICH E3 | SAC |
| Exposu | ire and Treatmo | ent Compliance | | | |
| 1.33. | Safety | EX1 | Summary of Exposure to Study Treatment: Part C | ICH E3 Dose and/or time on treatment, as applicable. | SAC |

# 10.11.5. Safety Tables

# 10.11.5.1. Safety Tables Part A

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events (AEs) | | | | |
| 2.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term: Part A | See Table 2.02 from 200975 | SAC |
| 2.2. | Safety | AE5a | Summary of All Adverse Events by System Organ Class and Maximum Intensity: Part A | ICH E3 | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | Safety | AE3 | Summary of Common (>10%) Adverse Events by Overall Frequency: Part A | GSK CTR | SAC |
| 2.4. | Safety | AE5a | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Intensity: Part A | GSK CTR | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 2.5. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class: Part A | IDSL / GSK CTR | SAC |
| 2.6. | Safety | AE3 | Summary of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency: Part A | IDSL | SAC |
| 2.7. | Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events: Part A | FDAAA, EudraCT | SAC |
| Labora | tory: Chemistry | <i>y</i> | | | |
| 2.8. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline: Part A | ICH E3 Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 2.9. | Safety | LB1 | Summary of Clinical Chemistry Values: Part A | | SAC |
| 2.10. | Safety | LB3 | Summary of Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part A | | SAC |
| 2.66. | Safety | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline: Part A | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hematolo | gy | | | |
| 2.11. | Safety | LB1 | Summary of Hematology Changes From Baseline: Part A | ICH E3 Includes baseline values. | SAC |
| 2.12. | Safety | LB1 | Summary of Hematology Values: Part A | ICH E3 Includes baseline values. | SAC |
| 2.13. | Safety | LB3 | Summary of Emergent Hematology Results by Potential Clinical Importance Criteria: Part A | | SAC |
| Labora | tory: Urinalysis | <b>5</b> | | <u> </u> | • |
| 2.14. | Safety | UR3 | Summary of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part A | ICH E3 Includes Baseline values. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | <u> </u> | • |
| 2.15. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting: Part A | IDSL | SAC |
| 2.16. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities: Part A | | SAC |
| ECG | | | | | |
| 2.17. | Safety | EG1 | Summary of ECG Findings: Part A | IDSL | SAC |
| 2.18. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit: Part A | IDSL | SAC |
| 2.19. | Safety | CP_EG12 | Summary of Maximum Change from Baseline in QTc Values by Category: Part A | IDSL | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | gns | | | | |
| 2.20. | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit: Part A | ICH E3<br>Includes Baseline values. | SAC |
| 2.21. | Safety | VS1 | Summary of Vital Signs by Visit: Part A | | SAC |

# 10.11.5.2. Safety Tables Part B

| Safety : | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.22. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term: Part B | See Table 2.02 from 200975 | SAC |
| 2.23. | Safety | AE5a | Summary of All Adverse Events by System Organ Class and Maximum Intensity: Part B | ICH E3 | SAC |
| 2.24. | Safety | AE3 | Summary of Common (>10%) Adverse Events by Overall Frequency: Part B | GSK CTR | SAC |
| 2.25. | Safety | AE5a | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Intensity: Part B | GSK CTR | SAC |
| Serious | Serious and Other Significant Adverse Events | | | | |
| 2.26. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class: Part B | IDSL / GSK CTR | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27. | Safety | AE3 | Summary of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency: Part B | IDSL | SAC |
| 2.28. | Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events: Part B | FDAAA, EudraCT | SAC |
| Labora | tory: Chemistry | / | | | |
| 2.29. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline: Part B | ICH E3 Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 2.30. | Safety | LB1 | Summary of Clinical Chemistry Values: Part B | | SAC |
| 2.31. | Safety | LB3 | Summary of Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part B | | SAC |
| 2.67. | Safety | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline: Part B | | SAC |
| Labora | tory: Hematolo | gy | | | |
| 2.32. | Safety | LB1 | Summary of Hematology Changes From Baseline: Part B | ICH E3 Includes baseline values. | SAC |
| 2.33. | Safety | LB1 | Summary of Hematology Values: Part B | ICH E3<br>Includes baseline values. | SAC |
| 2.34. | Safety | LB3 | Summary of Emergent Hematology Results by Potential Clinical Importance Criteria: Part B | | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Urinalysis | <b>.</b> | | | |
| 2.35. | Safety | UR3 | Summary of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part B | ICH E3<br>Includes Baseline values. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.36. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting: Part B | IDSL | SAC |
| 2.37. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities: Part B | | SAC |
| ECG | | | | | |
| 2.38. | Safety | EG1 | Summary of ECG Findings: Part B | IDSL | SAC |
| 2.39. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit: Part B | IDSL | SAC |
| 2.40. | Safety | CP_EG12 | Summary of Maximum Change from Baseline in QTc Values by Category: Part B | IDSL | SAC |
| Vital Si | gns | | | | |
| 2.41. | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit: Part B | ICH E3<br>Includes Baseline values. | SAC |
| 2.42. | Safety | VS1 | Summary of Vital Signs by Visit: Part B | | SAC |
| CSSRS | | | | | |
| 2.43. | Safety | CSSRS1 | Summary of Subjects with C-SSRS Suicidal Ideation or Behaviour during Treatment: Part B | | SAC |

# 10.11.5.3. Safety Tables Part C

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.44. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term: Part C | See Table 2.02 from 200975 | SAC |
| 2.45. | Safety | AE5a | Summary of All Adverse Events by System Organ Class and Maximum Intensity: Part C | ICH E3 | SAC |
| 2.46. | Safety | AE3 | Summary of Common (>10%) Adverse Events by Overall Frequency: Part C | GSK CTR | SAC |
| 2.47. | Safety | AE5a | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Intensity: Part C | GSK CTR | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 2.48. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class: Part C | IDSL / GSK CTR | SAC |
| 2.49. | Safety | AE3 | Summary of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency: Part C | IDSL | SAC |
| 2.50. | Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events: Part C | FDAAA, EudraCT | SAC |
| Labora | tory: Chemistry | / | | | • |
| 2.51. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline: Part C | ICH E3 Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 2.52. | Safety | LB1 | Summary of Clinical Chemistry Values: Part C | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.53. | Safety | LB3 | Summary of Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria: Part C | | SAC |
| 2.68. | Safety | LB17 | Summary of Worst Case Lipids Outside Laboratory Normal Range Post-Baseline Relative to Baseline: Part C | | SAC |
| Labora | tory: Hematolo | gy | | | |
| 2.54. | Safety | LB1 | Summary of Hematology Changes From Baseline: Part C | ICH E3 Includes baseline values. | SAC |
| 2.55. | Safety | LB1 | Summary of Hematology Values: Part C | ICH E3<br>Includes baseline values. | SAC |
| 2.56. | Safety | LB3 | Summary of Emergent Hematology Results by Potential Clinical Importance Criteria: Part C | | SAC |
| Labora | tory: Urinalysis | <b>5</b> | | | 1 |
| 2.57. | Safety | UR3 | Summary of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part C | ICH E3<br>Includes Baseline values. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.58. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting: Part C | IDSL | SAC |
| 2.59. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities: Part C | | SAC |
| ECG | | | | | |
| 2.60. | Safety | EG1 | Summary of ECG Findings: Part C | IDSL | SAC |
| 2.61. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit: Part C | IDSL | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.62. | Safety | CP_EG12 | Summary of Maximum Change from Baseline in QTc Values by Category: Part C | IDSL | SAC |
| Vital Sig | gns | | | | |
| 2.63. | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit: Part C | ICH E3 Includes Baseline values. | SAC |
| 2.64. | Safety | VS1 | Summary of Vital Signs by Visit: Part C | | SAC |

# 10.11.6. Safety Figures

# 10.11.6.1. Safety Figures Part A

| Safety : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.1. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk: Part A | IDSL | SAC |
| Hepato | bilary (Liver) | | | | |
| 2.2. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT: Part A | | SAC |
| 2.3. | Safety | LIVER9 | Scatter Plot for Maximum ALT va Maximum Total Bilirubin: Part A | | SAC |

# 10.11.6.2. Safety Figures Part B

| Safety : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.4. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk: Part B | IDSL | SAC |
| Hepato | bilary (Liver) | | | | |
| 2.5. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT: Part B | | SAC |
| 2.6. | Safety | LIVER9 | Scatter Plot for Maximum ALT va Maximum Total Bilirubin: Part C | | SAC |

# 10.11.6.3. Safety Figures Part C

| Safety : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.7. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk: Part C | IDSL | SAC |
| Hepato | bilary (Liver) | | | | |
| 2.8. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT: Part C | | SAC |
| 2.9. | Safety | LIVER9 | Scatter Plot for Maximum ALT va Maximum Total Bilirubin: Part C | | SAC |

## 10.11.7. Pharmacokinetic Tables

## 10.11.7.1. Pharmacokinetic Tables Part A

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 3.1. | PK | PK01 | Summary of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data by Formulation: Part A | Includes fed state. | SAC |
| PK Deri | ived Parameter | rs | | | |
| 3.2. | PK | PKPT1 | Summary Statistics of Derived Plasma GSK2982772 Pharmacokinetic Parameters by Formulation: Part A | Parameters with units. Includes fed state. | SAC |
| 3.3. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma GSK2982772 Pharmacokinetic Parameters by Formulation: Part A | Parameters with units. Includes fed state. | SAC |
| PK Ana | lyses | | | | |
| 3.4. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Formulation: Part A | | SAC |
| 3.5. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Formulation: Part A | Tmax | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Food Effect: Part A | | SAC |
| 3.7. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Food Effect: Part A | Tmax | SAC |
| 3.23. | PK | PK_T1 | Sensitivity: Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Formulation: Part A Excluding Subject | | SAC |
| 3.24. | PK | PK_T1 | Sensitivity: Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Formulation: Part A Excluding Subject | Tmax | SAC |
| 3.25. | PK | PK_T1 | Sensitivity: Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Food Effect: Part A Excluding Subject PPD | | SAC |
| 3.26. | PK | PK_T1 | Sensitivity: Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Food Effect: Part A Excluding Subject | Tmax | SAC |

## 10.11.7.2. Pharmacokinetic Tables Part B

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 3.8. | PK | PK01 | Summary of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data by Dose and Day: Part B | | SAC |
| PK Deri | ived Parameter | 'S | | | |
| 3.9. | PK | PKPT1 | Summary Statistics of Derived Plasma GSK2982772 Pharmacokinetic Parameters by Dose and Day: Part B | Parameters with units | SAC |
| 3.10. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma GSK2982772 Pharmacokinetic Parameters by Dose and Day: Part B | Parameters with units | SAC |
| 3.11. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2982772 Dose-Normalized Pharmacokinetic Parameters<br>by Dose and Day: Part B | Parameters with units | SAC |
| PK Ana | lyses | | | | |
| 3.12. | PK | PK_T2 | Summary of Statistical Analysis of Plasma GSK2982772 PK Parameters (AUC & C) Assessing Relative Bioavailability of Repeat Dose: Part B | | SAC |

## 10.11.7.3. Pharmacokinetic Tables Part C

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration | | | | |
| 3.13. | PK | PK01 | Summary of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data by Formulation/Prandial State: Part C | Includes fed state. | SAC |
| PK Der | ived Parameter | rs . | | | |
| 3.14. | PK | PKPT1 | Summary Statistics of Derived Plasma GSK2982772 Pharmacokinetic Parameters by Formulation/Prandial State: Part C | Parameters with units. Includes fed state. | SAC |
| 3.15. | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2982772 Pharmacokinetic Parameters by Formulation/<br>Prandial State: Part C | Parameters with units. Includes fed state. | SAC |
| 3.16. | PK | | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2982772 Dose-Normalized Pharmacokinetic Parameters by<br>Formulation/Prandial State: Part C | | |
| PK Ana | alyses | | | , | |
| 3.17. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Formulation: Part C | | SAC |
| 3.18. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Formulation: Part C | Tmax | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Food Effect: Part C | | SAC |
| 3.20. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Food Effect: Part C | Tmax | SAC |
| 3.21. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (AUC & C) Assessing Relative Bioavailability of Dose: Part C | | SAC |
| 3.22. | PK | PK_T1 | Summary of Statistical Analysis of Plasma GSK2982772 Parameters (Tmax) Assessing Relative Bioavailability of Dose: Part C | | SAC |

# 10.11.8. Pharmacokinetic Figures

# 10.11.8.1. Pharmacokinetic Figures Part A

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentrat | ion Plots | | | |
| 3.1. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time Plot by Subject (Linear and Semi-Log): Part A | Paginate by Subject | SAC |
| 3.2. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time Plot by Formulation (Linear and Semi-Log): Part A | Paginate by Formulation. This includes the fed state. | SAC |
| Mean / | Median Conce | ntration Plots | | | |
| 3.3. | PK | PKCF2 | Mean Plasma GSK2982772 Concentration-Time Plots by Formulation (Linear and Semi-log): Part A | Paginate by Formulation. This includes the fed state. | SAC |
| 3.4. | PK | PKCF3 | Median Plasma GSK2982772 Concentration-Time Plots by Formulation (Linear and Semi-log): Part A | Paginate by Formulation. This includes the fed state. | SAC |
| | 1 | 1 | | | 1 |
| 3.5. | PK | PK_F1 | Plot of Individual Subject (+Geometric Mean and 95% CI) Plasma GSK2982772 PK Parameters vs Formulation: Part A | | SAC |
| 3.6. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma GSK2982772 PK Parameters Assessing Relative Bioavailability of Formulation: Part A | | SAC |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.7. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Relative Bioavailability<br>of Food Effect: Part A | | SAC |

# 10.11.8.2. Pharmacokinetic Figures Part B

| Pharma | acokinetic: Figi | ıres | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentrat | ion Plots | | | |
| 3.8. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time Plot by Subject (Linear and Semi-Log): Part B | Paginate by Subject | SAC |
| 3.9. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time Plot by Dose (Linear and Semi-Log): Part B | Paginate by Dose | SAC |
| Mean / | Median Conce | ntration Plots | | | |
| 3.10. | PK | PKCF2 | Mean Plasma GSK2982772 Concentration-Time Plots by Dose (Linear and Semi-log): Part B | Paginate by Dose | SAC |
| 3.11. | PK | PKCF3 | Median Plasma GSK2982772 Concentration-Time Plots by Dose (Linear and Semi-log): Part B | Paginate by Dose | SAC |
| | 1 | | | | |
| 3.12. | PK | PK_F1 | Plot of Individual Subject (+Geometric Mean and 95% CI) Plasma GSK2982772 Dose-Normalized PK Parameters vs Dose: Part B | | SAC |
| 3.13. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Relative Bioavailability<br>of Repeat Dose: Part B | | SAC |

# 10.11.8.3. Pharmacokinetic Figures Part C

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentrati | on Plots | | | • |
| 3.14. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time Plot by Subject (Linear and Semi-Log): Part C | Paginate by Subject | SAC |
| 3.15. | PK | PKCF1P | Individual GSK2982772 Plasma Concentration-Time Plot by Formulation (Linear and Semi-Log): Part C | Paginate by Formulation. This includes the fed state. | SAC |
| Mean / | Median Conce | ntration Plots | | | • |
| 3.16. | PK | PKCF2 | Mean Plasma GSK2982772 Concentration-Time Plots by Formulation (Linear and Semi-log): Part C | Paginate by Formulation. This includes the fed state. | SAC |
| 3.17. | PK | PKCF3 | Median Plasma GSK2982772 Concentration-Time Plots by Formulation (Linear and Semi-log): Part C | Paginate by Formulation. This includes the fed state. | SAC |
| 3.18. | PK | PK_F1 | Plot of Individual Subject (+Geometric Mean and 95% CI) Plasma GSK2982772 PK Parameters vs Formulation: Part C | | SAC |
| 3.19. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma GSK2982772 PK Parameters Assessing Relative Bioavailability of Formulation: Part C | | SAC |
| 3.20. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Relative Bioavailability<br>of Food Effect: Part C | | SAC |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.21. | PK | PK_F2 | Plot of Geometric Mean Ratio and 90% CI of Plasma<br>GSK2982772 PK Parameters Assessing Relative Bioavailability<br>of Dose: Part C | | SAC |

# 10.11.9. ICH Listings

# 10.11.9.1. ICH Listing Part A

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |
| 1. | All Subjects | ES7 | Listing of Reasons for Screen Failure: Part A | Journal Guidelines | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal: Part A | ICH E3 | SAC |
| 3. | Safety | TA2 | Listing of Planned and Actual Treatments: Part A | IDSL | SAC |
| Protoc | ol Deviations | | | | 1 |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations: Part A | ICH E3 | SAC |
| 5. | All Subjects | IE4 | Listing of Subjectswith Inclusion/Exclusion Criteria Deviations: Part A | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | tions Analysed | | | | |
| 6. | Safety | SP3 | Listing of SubjectsExcluded from Any Population: Part A | ICH E3 | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | L |
| 7. | Safety | DM4 | Listing of Demographic Characteristics: Part A | ICH E3 | SAC |
| 8. | Safety | DM10 | Listing of Race: Part A | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 9. | Safety | CP_CM3 | Listing of Concomitant Medications: Part A | IDSL | SAC |
| Exposi | ure and Treatmo | ent Compliance | | | L |
| 10. | Safety | EX4 | Listing of Exposure Data: Part A | ICH E3 | SAC |
| Advers | se Events | | | | |
| 11. | Safety | AE9CP | Listing of All Adverse Events: Part A | ICH E3 | SAC |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events: Part A | ICH E3 | SAC |
| 13. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text: Part A | IDSL | SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 14. | Safety | AE9CP | Listing of Serious Adverse Events: Part A | ICH E3 | SAC |
| 15. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event: Part A | ICH E3 | SAC |
| ICH: Lis | ICH: Listings | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | | |
| 16. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment: Part A | ICH E3 | SAC | | | | |
| Hepato | biliary (Liver) | | | • | | | | | |
| 17. | Safety | MH2 | Listing of Medical Conditions for Subjectswith Liver Stopping Events: Part A | IDSL | SAC | | | | |
| 18. | Safety | SU2 | Listing of Substance Use for Subjectswith Liver Stopping Events: Part A | IDSL | SAC | | | | |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | |
| 19. | Safety | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range: Part A | ICH E3 | SAC |
| 20. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance: Part A | | SAC |
| 93. | Safety | LB6 | Listing of All Lipid Data for Subjects with Any Value Outside of Laboratory Normal Range: Part A | | SAC |
| 21. | Safety | LB14 | Listing of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part A | ICH E3 | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 22. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance: Part A | IDSL | SAC |
| 23. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance: Part A | IDSL | SAC |
| 24. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding: Part A | IDSL | SAC |
| 25. | Safety | EG6 | Listing of Abnormal ECG Findings: Part A | IDSL . | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | gns | | | | |
| 26. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance: Part A | IDSL | SAC |
| 27. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance: Part A | IDSL | SAC |

### 10.11.9.2. ICH Listings Part B

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | ct Disposition | | | | |
| 28. | All Subjects | ES7 | Listing of Reasons for Screen Failure: Part B | Journal Guidelines | SAC |
| 29. | Safety | ES3 | Listing of Reasons for Study Withdrawal: Part B | ICH E3 | SAC |
| 30. | Safety | TA2 | Listing of Planned and Actual Treatments: Part B | IDSL | SAC |
| Protoc | Protocol Deviations | | | | |
| 31. | Safety | DV2 | Listing of Important Protocol Deviations: Part B | ICH E3 | SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 32. | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations: Part B | ICH E3 | SAC |
| Popula | ations Analysed | | | | |
| 33. | Safety | SP3 | Listing of Subjects Excluded from Any Population: Part B | ICH E3 | SAC |
| Demog | graphic and Baseline | e Characteristics | 5 | | |
| 34. | Safety | DM4 | Listing of Demographic Characteristics: Part B | ICH E3 | SAC |
| 35. | Safety | DM10 | Listing of Race: Part B | ICH E3 | SAC |
| Prior a | and Concomitant Me | dications | | | |
| 36. | Safety | CP_CM3 | Listing of Concomitant Medications: Part B | IDSL | SAC |
| Expos | ure and Treatment C | Compliance | | | |
| 37. | Safety | EX4 | Listing of Exposure Data: Part B | ICH E3 | SAC |
| Advers | se Events | | | | |
| 38. | Safety | AE9CP | Listing of All Adverse Events: Part B | ICH E3 | SAC |
| 39. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events: Part B | ICH E3 | SAC |
| 40. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text: Part B | IDSL | SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Seriou | s and Other Signific | cant Adverse Eve | ents | • | |
| 41. | Safety | AE9CP | Listing of Serious Adverse Events: Part B | ICH E3 | SAC |
| 42. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event: Part B | ICH E3 | SAC |
| 43. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment: Part B | ICH E3 | SAC |
| Hepato | obiliary (Liver) | | | | |
| 44. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events: Part B | IDSL | SAC |
| 45. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events: Part B | IDSL | SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | |
| 46. | Safety | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range: Part B | ICH E3 | SAC |
| 47. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance: Part B | | SAC |
| 94. | Safety | LB6 | Listing of All Lipid Data for Subjects with Any Value Outside of Laboratory Normal Range: Part B | | SAC |
| 48. | Safety | LB14 | Listing of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part B | ICH E3 | SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 49. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance: Part B | IDSL | SAC |
| 50. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance: Part B | IDSL | SAC |
| 51. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding: Part B | IDSL | SAC |
| 52. | Safety | EG6 | Listing of Abnormal ECG Findings: Part B | IDSL | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital S | igns | | | | |
| 53. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance: Part B | IDSL | SAC |
| 54. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance: Part B | IDSL | SAC |
| C-SSR | S | • | | | |
| 55. | Safety | CSSRS4 | Listing of C-SSRS Suicidal Ideation and Behavior Data: Part B | IDSL | SAC |
| 56. | Safety | CSSRS5 | Listing of C-SSRS Suicidal Behavior Details: Part B | IDSL | SAC |
| PSRAE | PSRAE | | | | |
| 57. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data: Event and Description (Section 1 - Section 2): Part B | IDSL | SAC |

## 10.11.9.3. ICH Listing Part C

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | • | | | |
| 58. | All Subjects | ES7 | Listing of Reasons for Screen Failure: Part C | Journal Guidelines | SAC |
| 59. | Safety | ES3 | Listing of Reasons for Study Withdrawal: Part C | ICH E3 | SAC |
| 60. | Safety | TA2 | Listing of Planned and Actual Treatments: Part C | IDSL | SAC |
| Protoc | ol Deviations | 1 | | | 1 |
| 61. | Safety | DV2 | Listing of Important Protocol Deviations: Part C | ICH E3 | SAC |
| 62. | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations: Part C | ICH E3 | SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | ations Analysed | | | | |
| 63. | Safety | SP3 | Listing of Subjects Excluded from Any Population: Part C | ICH E3 | SAC |
| Demog | graphic and Baselin | e Characteristic | s | - | |
| 64. | Safety | DM4 | Listing of Demographic Characteristics: Part C | ICH E3 | SAC |
| 65. | Safety | DM10 | Listing of Race: Part C | ICH E3 | SAC |
| Prior a | nd Concomitant Me | dications | | | |
| 66. | Safety | CP_CM3 | Listing of Concomitant Medications: Part C | IDSL | SAC |
| Expos | ure and Treatment ( | Compliance | | 1 | - 1 |
| 67. | Safety | EX4 | Listing of Exposure Data: Part C | ICH E3 | SAC |
| Advers | se Events | | | • | |
| 68. | Safety | AE9CP | Listing of All Adverse Events: Part C | ICH E3 | SAC |
| 69. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events: Part C | ICH E3 | SAC |
| 70. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text: Part C | IDSL | SAC |
| Seriou | s and Other Signific | ant Adverse Eve | ents | | |
| 71. | Safety | AE9CP | Listing of Serious Adverse Events: Part C | ICH E3 | SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 72. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event: Part C | ICH E3 | SAC |
| 73. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment: Part C | ICH E3 | SAC |
| Hepato | Hepatobiliary (Liver) | | | | |
| 74. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events: Part C | IDSL | SAC |
| 75. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events: Part C | IDSL | SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | • | | | |
| 76. | Safety | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range: Part C | ICH E3 | SAC |
| 77. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance: Part C | | SAC |
| 95. | Safety | LB6 | Listing of All Lipid Data for Subjects with Any Value Outside of Laboratory Normal Range: Part C | | SAC |
| 78. | Safety | LB14 | Listing of Microscopy Results for Subjects with Abnormal Urinalysis Dipstick Results: Part C | ICH E3 | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 79. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance: Part C | IDSL | SAC |
| 80. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance: Part C | IDSL | SAC |
| 81. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding: Part C | IDSL | SAC |
| 82. | Safety | EG6 | Listing of Abnormal ECG Findings: Part C | IDSL | SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital S | Vital Signs | | | | |
| 83. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance: Part C | IDSL | SAC |
| 84. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance: Part C | IDSL | SAC |

# 10.11.10. Non-ICH Listings

### 10.11.10.1. Non-ICH Listings Part A

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | Pharmacokinetic | | | | |
| 85. | PK | PKCL1X | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-<br>Time (ng/mL) Data: Part A | | IA<br>SAC |
| 86. | PK | PKPL1X | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters: Part A | | IA<br>SAC |
| Meal Times | | | | | |
| 87. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days: Part A | | IA<br>SAC |

## 10.11.10.2. Non-ICH Listings Part B

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | Pharmacokinetic | | | | |
| 88. | PK | PKCL1 | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-<br>Time (ng/mL) Data: Part B | | IA<br>SAC |
| 89. | PK | PKPL1 | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters: Part B | | IA<br>SAC |

## 10.11.10.3. Non-ICH Listings Part C

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic | | | | |
| 90. | PK | PKCL1X | Listing of Plasma GSK2982772 Pharmacokinetic Concentration-<br>Time (ng/mL) Data: Part C | | IA<br>SAC |
| 91. | PK | PKPL1X | Listing of Derived Plasma GSK2982772 Pharmacokinetic Parameters: Part C | | IA<br>SAC |
| Meal Ti | Meal Times | | | | |
| 92. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days: Part C | | IA<br>SAC |